CLINICAL TRIAL: NCT02208310
Title: A Randomized Controlled Trial of High-Dose Vitamin D in Crohn's Disease
Brief Title: Trial of High Dose Vitamin D in Patient's With Crohn's Disease
Acronym: RODIN-CD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to enroll at rate anticipated, insufft low vitamin D in clin rem @ 5 sites
Sponsor: University of Michigan (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Peter Higgins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CCFA-329225
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-08

CONDITIONS: Crohn's Disease; Vitamin D Deficiency
Keywords: Crohn's disease; Vitamin D deficiency
MeSH Terms: conditions — Crohn Disease; Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Vitamin D (Active Comparator): Patients will be given 400 IU cholecalciferol once daily for 30 days. <-THIS IS THE Active Comparator Intervention. To maintain the blind, a random few will be given another round at the 30 day mark. For patients who enroll in the summer, a random few will again receive 400 IU cholecalciferol in March.
  Interventions: Drug: Cholecalciferol 400 IU
- High Dose Vitamin D (Experimental): Patients will be given cholecalciferol 10,000 IU daily for 30 days. <-THIS IS THE INTERVENTION. At that point, if their vitamin D levels remain below 50 ng/ml, the 30 day course will be repeated. For patients who enroll in the summer, levels will be rechecked in March and if <50 ng/ml, a 30 day course will be administered.
  Interventions: Drug: Cholecalciferol 10,000 IU

INTERVENTIONS:
Drug: Cholecalciferol 10,000 IU — Cholecalciferol 10,000 IU po daily
  Other Names: High Dose Vitamin D
  Arms: High Dose Vitamin D
Drug: Cholecalciferol 400 IU — Cholecalciferol 400 IU po daily
  Other Names: Low dose vitamin D
  Arms: Low Dose Vitamin D

SUMMARY:
Crohn's disease is more common in areas of the world with less sunlight exposure. Sunlight is a major source of vitamin D. There is some research to suggest that patient's with higher vitamin D levels are less likely to undergo surgeries and have better control of their disease. We intend to study the effects of high dose vitamin D supplementation in patients with vitamin D deficiency and Crohn's disease. We hypothesize that patients given high doses will have less hospitalizations, surgeries, steroid use.

DETAILED DESCRIPTION:
Subjects are randomized to low or high dose vitamin D, and outcomes including steroid prescriptions, CD-related hospitalizations, CD-related surgeries, and the modified Harvey-Bradshaw Index are measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD
* Age >= 18 and <75
* Vitamin D deficiency or insufficiency (serum 25-hydroxyvitamin D < 30ng/ml)

Exclusion Criteria:

* Corticosteroid use in the last 4 weeks
* CD-related surgery in the last 6 months
* CD-related hospitalization in the last 4 weeks
* Pregnancy, intended pregnancy during the study period or nursing
* Serum calcium >10.2 mg/dL
* History of primary sclerosing cholangitis
* History of undergoing an ileal pouch-anal anastomosis
* Current active perianal disease
* History of nephrolithiasis in the past 2 years
* Anticipated change in therapy in the next 30 days (steroids, biologic initiation)
* modified Harvey-Bradshaw Index of 10 or more
* History of decreased renal function (glomerular filtration rate <30ml/min based on MDRD) or polycystic kidney disease
* History of sarcoidosis
* History of hyperparathyroidism
* Any other chronic condition that may preclude high doses of Vitamin D such as lymphoma
* Concurrent use of hydrochlorothiazide, phenytoin, phenobarbital, carbamazepine or primidone
* Osteoporosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter D. Higgins, MD, PhD, MSc, Principal Investigator — University of Michigan; Shail M Govani, M.D., M.Sc., Study Director — University of Michigan; Hans Herfarth, MD, PhD, Study Director — University of North Carolina
Locations (4):
- United States (4):
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- [Background] Jorgensen SP, Agnholt J, Glerup H, Lyhne S, Villadsen GE, Hvas CL, Bartels LE, Kelsen J, Christensen LA, Dahlerup JF. Clinical trial: vitamin D3 treatment in Crohn's disease - a randomized double-blind placebo-controlled study. Aliment Pharmacol Ther. 2010 Aug;32(3):377-83. doi: 10.1111/j.1365-2036.2010.04355.x. Epub 2010 May 11. PMID 20491740
- [Background] Khalili H, Huang ES, Ananthakrishnan AN, Higuchi L, Richter JM, Fuchs CS, Chan AT. Geographical variation and incidence of inflammatory bowel disease among US women. Gut. 2012 Dec;61(12):1686-92. doi: 10.1136/gutjnl-2011-301574. Epub 2012 Jan 11. PMID 22241842
- [Background] Cantorna MT, Munsick C, Bemiss C, Mahon BD. 1,25-Dihydroxycholecalciferol prevents and ameliorates symptoms of experimental murine inflammatory bowel disease. J Nutr. 2000 Nov;130(11):2648-52. doi: 10.1093/jn/130.11.2648. PMID 11053501
- [Background] Ananthakrishnan AN, Khalili H, Higuchi LM, Bao Y, Korzenik JR, Giovannucci EL, Richter JM, Fuchs CS, Chan AT. Higher predicted vitamin D status is associated with reduced risk of Crohn's disease. Gastroenterology. 2012 Mar;142(3):482-9. doi: 10.1053/j.gastro.2011.11.040. Epub 2011 Dec 9. PMID 22155183

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Vitamin D: Patients will be given 400 IU cholecalciferol once daily for 30 days. To maintain the blind, a random few will be given another round at the 30 day mark. For patients who enroll in the summer, a random few will again receive 400 IU cholecalciferol in March.
  Cholecalciferol 400 IU
- High Dose Vitamin D: Patients will be given cholecalciferol 10,000 IU daily for 30 days. At that point, if their vitamin D levels remain below 50 ng/ml, the 30 day course will be repeated. For patients who enroll in the summer, levels will be rechecked in March and if <50 ng/ml, a 30 day course will be administered.
  Cholecalciferol 10,000 IU
Period: Overall Study
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Started | 6 | 5
Day 180 | 0 | 1
Completed | 0 | 0
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (14.2) | 35.2 (9.0) | 34.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint: Number of Participants With (Any of) a CD-related Hospitalization, CD-related Surgery, CD-related ER Visits and Steroid Prescriptions
Description: Composite endpoint of (any of) Crohn's disease(CD)-related hospitalizations, CD-related surgeries, CD-related ER visits, or steroid prescriptions.
  Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Number; unit: participants
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
participants |  | 0

2. Primary Outcome: Hypercalcemia
Description: Hypercalcemia is presented as number of participants with Calcium >10.8 mg/dl Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
Participants |  | 0

3. Primary Outcome: Incidence of Nephrolithiasis
Description: Incidence of nephrolithiasis associated with hypercalcemia (>10.8mg/dl) documented by imaging Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
Participants |  | 0

4. Secondary Outcome: Crohn's Related Hospitalizations
Description: Dichotomous (0/1) endpoint for each subject, depending on whether a CD-related hospitalization occurred. Relatedness to Crohn's disease as judged by the DSMB. Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Number; unit: CD-related hospitalization occurred
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
CD-related hospitalization occurred |  | 0

5. Secondary Outcome: Steroid Prescription Given (Dichotomous 0/1)
Description: Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here. No steroid prescriptions occurred
Time Frame: Day 180
Measure: Number; unit: Steroid prescription occurred
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
Steroid prescription occurred |  | 0

6. Secondary Outcome: Crohn's Related Surgeries (Dichotomous 0/1 Per Subject)
Description: Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here. No CD-related surgeries occurred in the 1 subject
Time Frame: Day 180
Measure: Number; unit: CD-related surgery occurred
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
CD-related surgery occurred |  | 0

7. Secondary Outcome: Change in Modified Harvey-Bradshaw Index (HBI Without Examination)
Description: modified Harvey-Bradshaw is a disease assessment scale. 0 is the lowest score and would be considered remission. Scale ranges to over 16 (upper limit is defined by the number of bowel movements in the prior day) with numbers over 16 being severe disease. A positive change (such as that indicated below) therefore references slightly worsening disease while a negative change references improving disease.
  Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here. 1 subject had an increase of 1 unit on the modified HBI.
Time Frame: Day 180
Measure: Number; unit: units on a scale (0-16)
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
units on a scale (0-16) |  | 1

8. Secondary Outcome: Change in C-reactive Protein
Description: Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here. The delta between first (baseline) and last CRP (Day 180) is reported here.
Time Frame: Day 180
Measure: Number; unit: mg/dL
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
mg/dL |  | 0

9. Secondary Outcome: Changes in Fecal Calprotectin
Description: Originally planned to collect at Day 180 and Day 360. Results were not collected on any subjects, as the one participant did not provide a stool sample.
Time Frame: 1 year
Population: Results were not collected on any subjects
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percent With Escalation of Therapy
Description: Patients who had to have a change in therapy Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
Participants |  | 0

11. Secondary Outcome: Quality of Life Measure Changes
Description: change in quality of life measures based on Inflammatory bowel disease questionnaire (IBD-Q).
  Scale from 0 to 224 with 0 being the poorest quality of life and 224 being the highest quality of life. A positive change indicates improvement while a negative change indicates worsening.
  Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Number; unit: units on a scale
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
units on a scale |  | -7

12. Secondary Outcome: Change in Fatigue Measurements
Description: Change in FACIT-F scale over the year. Scale is 0-160 with 0 being no fatigue and 160 being extreme fatigue. A positive change indicates worsening in symptoms and a negative change indicates an improvement.
  Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here.
Time Frame: Day 180
Measure: Number; unit: units on a scale
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
units on a scale |  | -3

13. Secondary Outcome: Participants With at Least One Crohn's Related Emergency Department (ED) Visit
Description: Originally planned to collect at Day 180 and Day 360. Only 1 subject remained in the study to Day 180 so that data is presented here. No CD-related ED visits occurred in the 1 subject
Time Frame: Day 180
Measure: Number; unit: participants
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
Number analyzed (Participants) | 0 | 1
participants |  | 0

ADVERSE EVENTS:
Time Frame: AEs are reported for as long as participants remained in the study. All but one had left short of 6 months; one continued through the 6 month milestone.
Description: Not different
Arm/Group | Low Dose Vitamin D | High Dose Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Vitamin D (N=6) | High Dose Vitamin D (N=5)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Urinary Tract Infection

LIMITATIONS AND CAVEATS:
Very few patients with inactive disease had low vitamin D levels, so most patients screened were ineligible. This made recruitment very slow, and the project was terminated.Suggests low vitamin D could be a marker of activity, rather than a cause

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No